CLINICAL TRIAL: NCT04645706
Title: Innate T-cells as a Biomarker of Successful TKI Arrest in Chronic Myeloid Leukemia
Brief Title: Innate T Cells and TKI Discontinuation
Acronym: TIBIOP-LMC
Status: Active, not recruiting | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TIBIOP-LMC
Record Dates: First submitted 2020-05-06; First posted 2020-11-27 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Characteristics of innate T cells — functional and phenotypic characteristics of innate T cells

SUMMARY:
After more than a decade of treating chronic myeloid leukemia (CML) with tyrosine kinase inhibitors (TKI), the discontinuation of treatment represents the expected new revolution. The investigators has recently discovered a new innate CD8+ T population in healthy subjects, the Eomes+ KIR+ CD8+ T population, with anti-tumor properties. Remarkably, these cells are numerically and functionally deficient in patients at diagnosis and then restored in patients in major molecular remission (MMR) on TKI. Our work performed in a retrospective pilot study interestingly shows a very significant increase in the proportion of CD8+ Eomes+ KIR+ T cells within total T cells in patients with prolonged success in stopping their ITK (≥ 2 years).Thus, the investigators postulate that CD8+ Eomes+ KIR+ T cells are a predictive signature of TKI arrest success in CML. The investigators will rely on a prospective translational study of this cell contingent during treatment cessation.

DETAILED DESCRIPTION:
To perform this research, the investigators have started a prospective translational study to collect samples in CML patients with successful versus patients who have failed TKI therapy discontinuation. The investigators plan to study functional and phenotypic characteristics of innate T cells. The investigators also plan to evaluate in vitro whether immune check points inhibitors could help to restore the innate T lymphocytes population.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Diagnosis of CML-PC according to the criteria of the European Leukemia Net (Baccarani et al, 2013)
* Patients treated with TKI for at least 3 years (imatinib, nilotinib, dasatinib, bosutinib, ponatinib)
* Patients meeting the criteria of the French STIM study: deep molecular response of MR4.5 type (threshold of 0.0032%) or MR5 type (threshold of 0.001%) for at least 2 years,
* Free subject, without guardianship or curatorship or subordination
* Patients benefiting from a Social Security system or benefiting from it through a third party

Exclusion Criteria:

* Refusal to participate in the research
* Patients not benefiting from a Social Security scheme or not benefiting from it through a third party
* Persons benefiting from enhanced protection, namely minors, persons deprived of their liberty by a judicial or administrative decision, persons staying in a health or social institution, adults under legal protection, and finally patients in emergencies
* Patient having stopped treatment for another reason than: deep molecular response of MR4.5 (threshold of 0.0032%) or MR5 (threshold of 0.001%) for at least 2 years

Translated with www.DeepL.com/Translator (free version)

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: CML patients for whom treatment with TKI is stopped according to the recommendations of the French Fi-LMC group.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Compare the quantitative characteristics of the CD8+ Eomes+ KIR+ T cells between patients in failure versus those in success after discontinuation of TKI treatment | Day 0 (day of discontinuing treatment)
  Proportion of the CD8+ Eomes+ KIR+ T cells among CD8+ T cells between patients in failure versus those in success after discontinuation of TKI treatment
Compare phenotypic characteristics of the CD8+ Eomes+ KIR+ T cells between patients in failure versus those in success after discontinuation of TKI treatment | Day 0 (day of discontinuing treatment)
  Phenotypic markers expression : CD49d, CD57, CD45RA et CCR7, CD25 et HLA-DR among total CD8+ T cells
Compare the functionnality of the CD8+ Eomes+ KIR+ T cells between patients in failure versus those in success after discontinuation of TKI treatment | Day 0 (day of discontinuing treatment)
  Functionality of LT CD8+ Eome+ KIR+ : expression of perforin and IFNgamma

CONTACTS AND LOCATIONS:
Overall Officials: Emilie CAYSSIALS, Study Director — Poitiers University Hospital
Locations (1):
- C.H.U. de Poitiers, Poitiers, France